CLINICAL TRIAL: NCT01504542
Title: A Phase 2A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Immune Response, Safety and Efficacy of HS-110 in Combination With Erlotinib vs. Erlotinib as a Single Agent in Patients With Advanced, Non-EGFR Mutated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Immune Response and Safety of HS110 Vaccine in Combination With Erlotinib in Patients With Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Heat Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS110-10-01
Record Dates: First submitted 2011-12-20; First posted 2012-01-05 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low-dose HS-110 (Experimental): 2,000,000 cells/0.5mls + erlotinib 150mg orally once daily
  Interventions: Biological: HS110 vaccine
- High dose HS110 (Experimental): 10,000,000 HS110 cells/0.5ml + erlotinib 150mg orally once daily.
  Interventions: Biological: HS110 vaccine
- Placebo vaccine + erlotinib 150mg orally once daily (Placebo Comparator): Placebo vaccine buffered saline solution + erlotinib 150mg orally once daily
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HS110 vaccine — 0.5ml to be administered twice weekly for 18 weeks (36 doses)
  Arms: Low-dose HS-110
Biological: Placebo — 0.5ml buffered saline placebo to be administered twice weekly for 18 weeks (36 doses)
  Arms: Placebo vaccine + erlotinib 150mg orally once daily
Biological: HS110 vaccine — 0.5 mls to be dosed twice weekly for 18 weeks (36 doses)
  Arms: High dose HS110

SUMMARY:
This study will enroll patients with locally advanced or metastatic non-EGFR mutated Non-Small Cell Lung Cancer (NSCLC) lung cancer after failure of at least one but no more than two prior approved treatment regimens. Patients will be randomized to receive one of two doses of vaccine or placebo to be dosed twice weekly for 18 weeks (36 doses total) and patients will also receive erlotinib 150mg taken orally once daily for the duration of the trial. The study will examine the immune effects, safety and efficacy of two different doses of HS110 vaccine in combination with erlotinib versus erlotinib alone.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled study will enroll patients with advanced NSCLC (squamous cell or non-squamous cell) without EGFR mutations (either L858R or 746-750 deletions) who have had progression or recurrence of their disease following at least one but no more than two prior regimens (adjuvant therapy excluded) of approved therapy that did not include immunomodulating or anti-EGFR targeted therapy for their disease. EFGR status must be known at the time of enrollment either via prior determination or testing performed from archival tissue during the screening process. Patients with resectable disease will eligible if resection can be deferred for the first six weeks of vaccine. Patients will receive twice weekly dosing of vaccine (spatially divided as 5 intradermal injections) for 18 weeks (36 total doses). Patients will be randomized in a 2:1 fashion; with 30 patients in each of the HS110 treatments groups (high and low dose) and 15 patients will receive placebo injections. Patients will also receive erlotinib 150mg once daily for the duration of the trial. A total of 75 patients will be enrolled in the trial. The study includes a lead-in phase of 9 patients (3 from each dosing group) who will be observed weekly for 4 weeks to assess the safety of combining HS110 with erlotinib. Treatment of the first 4 patients will be staggered by 2 week intervals to allow for safety evaluation before treating additional patients. If the combination of proves to be safe and well-tolerated in the first 9 patients, enrollment will be opened up to the predetermined sample size for each arm. A Data Monitoring Committee (DMC) will be used in this study to independently monitor adverse events and progression/survival data. The DMC will meet at the completion of the run-in period and after half the patients have been dosed through week 6 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with the protocol and sign informed consent.
* Histologically or cytologically confirmed locally advanced or metastatic squamous cell or non-squamous cell NSCLC after at least one but no more than two prior regimens of approved therapy for their disease (not including adjuvant treatment).
* Confirmation that their disease has no known EGFR mutations based on documented prior analysis or study-specific analysis of archival tumor tissue.
* At least one site of bi-dimensionally measurable NSCLC disease.
* Patients with recurrent, resectable disease able to undergo six weeks of vaccine therapy prior to resection.
* Brain metastasis if present and treated must be stable by CT scn or MRI for at least 8 weeks.
* Age ≥ 18 years.
* EGOG performance status of 0-1.
* Lab parameters
* Albumin ≥ 3.5mg/dL
* Total Bilirubin < 1.5mg/dL
* Alanine transaminase (ALT), and aspartate transaminase(AST)≤ 2.5 x upper limits of normal or ≤ x ULN in case of liver metastases.
* Serum creatinine < 1.5mg/dL or calculated creatinine clearance >50 mL/minute per the Cockcroft-Gault formula.
* White blood cell (WBC) count ≥ 4,000/mm3 with an absolute neutrophil count

  * 1,500mm3.
* Hemoglobin ≥ 9g/dL
* Platelet count ≥ 100,000/mm3
* Women of childbearing potential or men of fathering potential must use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide or surgical sterilization) during the study and for 6 months after receiving the last administration of study medication. Female patients of childbearing potential must test negative for pregnancy prior to enrolling in the trial. Post-menopausal (cessation of menses for more than 6 months) women are eligible for this study.

Exclusion Criteria:

* No prior therapy with EGFR-targeted drugs, including approved and investigational therapies, or prior immunologic or biologic response modifier therapy for treatment of their disease.
* Uncontrolled or untreated brain or spinal cord metastases or meningeal carcinomatosis.
* Known human immunodeficiency virus (HIV), hepatitis B or C, or severe/uncontrolled infections or intercurrent illness, unrelated to the tumor, requiring active therapy.
* Autoimmunity syndromes (primary or acquired) including, but not limited to, the following: rheumatoid arthritis, systemic lupus erythematosus, Sjogren's disease, sarcoidosis, vasculitis, polymyositis, or glomerulonephritis requiring active steroid or other immunosuppressive therapy.
* Known immunodeficiency disorders, either primary or acquired.
* Other malignancies present within the past 3 years, except for cutaneous basal and/or squamous cell carcinoma(s) or in situ cervical cancer.
* History of clinically significant cardiac impairment, congestive heart failure > New York Heart Association (NYHA) cardiac disease classification Class II, unstable angina, or myocardial infarction during the previous 6 months, or serious cardiac arrhythmia.
* Known alcohol or chemical abuse, or mental or psychiatric condition precluding compliance with the protocol.
* Chemotherapy, radiation, or other antitumor therapy during the last 4 weeks.
* Pregnant, nursing, or planning a pregnancy (both men and women) within 12 months of enrollment.
* Known allergy to soy or egg products.
* Patient is anaplastic lymphoma kinase (ALK)-positive as detected by an FDA-approved test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Immunologic Response (defined as production of IFNƴ from CD8+ T cells as evaluated by ELISPOT assay) | Week 18
  Immune response will be evalulated by ELISPOT assays and change will be assessed from baseline.

SECONDARY OUTCOMES:
Safety of the combination of HS110 vaccine and erlotinib | Up to 1 year
  Incidence and severity of adverse events, changes in laboratory measures, physical exams and evaluation of autoimmune phenomena.
Tumor assessment by immunologic response criteria (irRC) | Baseline, Week 12 and Week 22
  Patients will have a CT scan performed at baseline, Week 12 and Week 22 or at the end of study visit in the case of early termination from study. Investigators will assess the disease response using irRC for overall response, CR, PR, SD or PD.
Exploratory Immunologic endpoint - evaluation of circulating tumor cells | Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12 and Week 18
  Analysis via a semiautomated, epithelial cell adhesion molecule-based immunomagnetic technique.
Exploratory immunologic endpoint - immune function | Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12 and Week 18
  Analysis of cell surfance molecules by flow cytometry
Exploratory immunologic endpoint - proteomic profile | Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 9, Week 12 and Week 18
  Examination of protein expression utilizing western blot, immunohistochemical staining, enzyme linked immunosorbent assay (ELISA) or mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Principal Investigator — Mary Crowley Cancer Research Centers
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States